CLINICAL TRIAL: NCT03523806
Title: Children and Teens in Charge of Their Health: A Feasibility Study of Solution-focused Coaching to Foster Healthy Lifestyles in Children and Young People With Physical Disabilities
Brief Title: Children and Teens in Charge of Their Health
Acronym: CATCH
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Holland Bloorview Kids Rehabilitation Hospital (Other)
Collaborators: Laval University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: CATCH-17-752
Record Dates: First submitted 2018-04-12; First posted 2018-05-14 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Spina Bifida; Cerebral Palsy; Health Behavior
MeSH Terms: conditions — Spinal Dysraphism; Cerebral Palsy; Health Behavior

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Solution-Focused Coaching Group (Experimental): Half of the participants (n=15) will be assigned a coach and receive coaching 8 times for up to 1 hour over 6 months. The first session will take place in the home and subsequent session will take place online using an online meeting tool.
  Interventions: Behavioral: Solution-Focused Coaching in Pediatric Rehabilitation
- Control Group (No Intervention): Half of the participants (n=15) will not be receiving coaching

INTERVENTIONS:
Behavioral: Solution-Focused Coaching in Pediatric Rehabilitation — A coaching model for children with disabilities, with a strong theoretical basis, and ability to be customized to children and families' resources, environmental settings, child age and developmental stage
  Arms: Solution-Focused Coaching Group

SUMMARY:
This three year study explores the feasibility and acceptability of conducting a full randomized controlled trial (RCT) of a promising coaching intervention for improving and sustaining physical activity (PA) and healthy dietary habits in children with physical disabilities (CWPD).

Thirty children (ages 10 - 18) will spend 12 months in the study. All will receive usual care and basic printed information about healthy lifestyles. In addition, 15 will receive a coaching intervention for the first six months. Pre-defined success criteria will assess the feasibility of trial processes.

Acceptability of trial participation and impact of coaching will be explored qualitatively. Health indicators and psychosocial outcomes will be assessed four times, at the start of the trial, immediately post-intervention and at three and six months post-intervention.

DETAILED DESCRIPTION:
The World Health Organization's Global Strategy on Diet, Physical Activity (PA) and Health Promotion highlights that PA and dietary habits are central to disease prevention and lifelong health. Canadian children have increased health risks as their activity levels are drastically lower than recommendations and ~26% are classified as overweight or obese. The situation is even more critical for children with disabilities; 4.2% of Canadian children have disabilities and this number is rising. Due to complex and intersecting factors, children with physical disabilities (CWPD) are more sedentary, have lower PA rates and poorer quality diets than their non-disabled peers. Annual health care costs of obesity related to disability are estimated at $44 billion in the US, supporting the need to start health promotion activities early in life. Despite the serious proximal and distal consequences of this health profile, the investigators lack robust evidence on effective strategies to foster and sustain health habits for CWPD.

A new intervention paradigm that produces sustainable results without undue burden (on families or services) is therefore urgently required to address the health promotion needs of CWPD. The investigators propose that a strengths-based coaching approach may meet all of these requirements. Solution-Focused Coaching in Pediatric Rehabilitation (SFC-Peds) has been recommended as a coaching model for children with disabilities, for its strong theoretical basis and ability to be customized to children and families' resources, environmental settings, child age and developmental stage. Taking a strengths-based approach (such as SFC-Peds) is a departure from usual rehabilitation research and practice, which has largely been problem-focused (i.e. what a child can't do). A strengths-based approach can result in hope, motivation and action.

Given that the investigators will be the first to use SFC-Peds to promote healthy habits with CWPD, a feasibility and acceptability study is essential. Evidence of feasibility is a critical prerequisite for a RCT, especially for complex interventions that have multiple interacting components and/or target multiple behaviours (such as SFC-Peds). Feasibility studies rigorously examine the processes (e.g. recruitment and retention), resources (e.g. personnel, time required to complete measures), management (e.g. coordination of research personnel, quality of data entry) and science (e.g. appropriate methodology and outcomes) of the intended RCT. It is also critical to evaluate the acceptability of interventions for the target population (e.g. satisfaction with duration, intensity, level of interest, perceived impact), as well as those allocated to the control arm (e.g. acceptability of not receiving coaching, perceived burden of assessments). Examining all of these issues before the efficacy trial begins increases the likelihood of success. Feasibility studies such as the one the investigators are proposing help ensure that resources are invested in efficacy trials likely to generate clinically meaningful results and therefore have maximum impact on health care knowledge and outcomes.

Primary objective: To evaluate the feasibility (study design, methods, processes) and acceptability (family/child/clinician satisfaction, perceived usefulness) of conducting a randomized controlled trial (RCT) of a novel, brief, coaching intervention, solution-focused coaching in pediatric rehabilitation (SFC-Peds) for improving and sustaining physical activity (PA) and dietary habits in children with physical disabilities (CWPD).

Secondary objective: To determine the responsiveness of selected outcome measures to SFC-Peds coaching over 12 months.

Principal research question: "Is an efficacy trial to evaluate a 6 month SFC-Peds intervention to improve PA and dietary habits feasible to implement and acceptable to CWPD and families?"

Physical, environmental and psychosocial restrictions mean that children with physical disabilities (CWPD) are adopting worrying physical activity (PA) and dietary habits. Despite this, the investigators currently have limited evidence to inform interventions that may enhance lifelong health in CWPD. The investigators suggest that a paradigm shift is needed, one that moves beyond traditional prescriptive programs to a strengths-based approach where intervention strategies enable new health habits to be integrated seamlessly into children and families' everyday lifestyles for long-term sustainability.

Research such as our proposed study will ensure that this potentially transformative approach is rigorously examined and used in an evidence-based manner. As little is known about effective and acceptable behaviour change interventions for CWPD, this study's findings will make significant contributions to the field: i) Greater understanding of ecologically valid interventions that have the potential to enhance the long term health of CWPD; ii) Insight into how 2 different rehabilitation populations respond to SFC-Peds; and iii) Data on the responsiveness of outcome measures to a SFC-Peds intervention. These insights will enable us to design acceptable, feasible and rigorous interventions that will result in robust data for informing both research and clinical practice.

ELIGIBILITY:
Child Inclusion Criteria:

* Between the age of 10 - 18 years inclusive
* Diagnosis of SB or CP
* Has physical capability to execute independent body movement with or without device
* Cognitively able and willing to set PA or dietary goals
* Can communicate in English and respond to questions requiring some reflection and insight
* Home internet connection
* Lives within 2 hours driving distance from Toronto up to London, Ontario OR willing to travel to either HB or TVCC for first in-person coaching session if randomized into coaching group

Child exclusion criteria:

* Surgery in past 6 months or upcoming 12 months that may impact PA or dietary intake (e.g. orthopedic surgery or neurosurgery)
* Medical condition severely restricting diet
* Underweight (less than fifth percentile)
* Receiving specialist dietetic services

Parent inclusion criteria:

* Primary caregiver to a study participant
* Can communicate in English and respond to questions requiring some reflection and insight

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 16 (Actual)
Dates: Start 2018-03-23 (Actual); Primary Completion 2023-03-31 (Estimated); Study Completion 2023-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) scores | At first coaching session (immediately post-study enrollment/randomization) and at Time 2 (immediately post-coaching), 3 (3 months post-coaching), 4 (6 months post-coaching)
  The COPM is an evidence-based outcome measure designed to capture a participant's self-perception of performance in everyday living, over time.
  Participants will identify occupational performance problems in the areas of SELF-CARE (personal care, functional mobility, and community management), PRODUCTIVITY (paid or unpaid work, household management, and school and/or play), and LEISURE (quiet recreation, active recreation, and socialization).
  They will then rate each one in terms of its IMPORTANCE in their life on a scale of 1 (not important at all) to 10 (extremely important). Respondents will pick 5 problems and for each problem rate:
  PERFORMANCE (how would you rate the way that you do this activity now?) on a scale of 1 (not able to do it at all) to 10 (able to do it extremely well) SATISFACTION (How satisfied are you with the way you do this activity now?) on a scale of 1 (not satisfied at all) to 10 (extremely satisfied).

SECONDARY OUTCOMES:
Change Goal Attainment Scaling (GAS) scores | At first coaching session (immediately post-study enrollment/randomization) and at Time 2 (immediately post-coaching), 3 (3 months post-coaching), 4 (6 months post-coaching)
  A measure of participant goal attainment by defining five levels of goal attainment, thus ensuring that all attainment levels are mutually exclusive and measurable. This is an objective measure of behaviour change. Participants will provide a goal statement for each level.
  Scale ranges from:
  * 2 present level or much less than expected
  * 1 somewhat less than expected 0 expected level or program goal
    * 1 somewhat better than expected
    * 2 much better than expected A single GAS score is identified for a goal from the above 5 levels. Higher scores indicate better goal attainment.

OTHER OUTCOMES:
Change in Habitual Activity Estimation Scale scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  A child questionnaire estimating percent of time spent inactive, somewhat inactive, somewhat active, and very active on a typical school day and Saturday. Each question represents 1 time point in the day. Estimated percent ranging from 0-100% for all 4 activity levels must add up to 100% per question.
  Activity Level Description
  * Inactive - lying down, resting
  * Somewhat inactive - activities that are mostly done sitting down.
  * Somewhat active - walking, shopping, light chores, playing with pet
  * Very active - require lots of movement and make you breathe/sweat hard
  The questionnaire also asks participants to rate their:
  * Overall level of activity (very inactive to very active) on a typical school day/Saturday
  * How typical the school day/Saturday described was in the last 6 months (very much like most days to very different from most days)
  * Changes in a participant's activity level from 6 months on a school day/weekend (choice of much less active to much more active)
Change in Dietary Screener Questionnaire scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  A child questionnaire assessing dietary intake over the past 30 days and is validated against 24 hour multiple recall.
  The questionnaire asks participants they had specific types of foods and beverages in the last month as well as the type of milk and cereals consumed.
  For beverages, the scale ranges are:
  * Never
  * 1 time last month
  * 2 - 3 times last month
  * 1 time per week
  * 2 times per week
  * 3 - 4 times per week
  * 5 - 6 times per week
  * 1 time per day
  * 2 - 3 times per day
  * 6 or more times per day
  For food, the scale ranges are:
  * Never
  * 1 time last month
  * 2 - 3 times last month
  * 1 time per week
  * 2 times per week
  * 3 - 4 times per week
  * 5 - 6 times per week
  * 1 time per day
  * 2 or more times per day
Change in Arc's Self-Determination Scale scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  A child questionnaire assessing self-determination. Only multiple choice domains 1 (autonomy), 3 (psychological empowerment), and 4 (self-realization) will used.
  Domain 1 scores range from 0 ("I don't even have a chance) to 3 (I do every time I have a chance) for each question (21 questions) and summed (max. score of 96). Higher scores indicate higher levels or autonomy.
  Domain 2 scores are 0 or 1 (16 points total) depending on response. Answers reflecting psychological empowerment (e.g. beliefs in ability, perceptions of control, and expectations of success) are scored 1 and those that do not reflect a psychologically empowered belief or attitude are scored 0. Higher scores indicate more psychological empowerment.
  Domain 3 scores are 0 (answer not reflecting positive self-awareness/knowledge) or 1 (answer reflecting positive self-awareness/knowledge) based on response (total 15 points). Higher scores represent greater self-realization.
Change in Physical Activity Self-efficacy Scale scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  A child questionnaire assessing confidence in the ability to be physically active when faced with challenges. Participants will rate each physical activity self-efficacy statement with either a "yes" or "no" (e.g. I think I can ask my parents or another adult to sign me up for a physical activity - yes or no?). Higher number of "yes" responses indicate higher physical activity self-efficacy.
Change in Self-Efficacy for Healthy Eating scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  A child questionnaire assessing participants' feelings of competence for making healthy food choices in: social, emotional, and typical situations.
  Participants rate each self-efficacy statement for healthy eating (e.g. If you wanted to, how sure are you that you could eat healthy foods when you are… at the mall.. with your friends..etc.) on a scale ranging from:
  * Not sure at all
  * Not sure
  * Neither sure nor unsure
  * Fairly sure
  * Very sure Higher scores indicate higher self-efficacy for healthy eating.
Change in BMI | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  Weight will be measured in kg and height will be measured in cm to determine BMI calculated based on height and weight in kg/m^2
Change in the Family Eating and Activity Habits Questionnaire scores | Time 1 Baseline (upon study enrollment), Time 2 (6 months post-baseline or immediately post-coaching), 3 (9 months post-baseline or 3 months post coaching), 4 (12 months post-baseline or 6 months post-coaching)
  This is a 32-item parent-report assessment to assess the health behaviours of family members as well as the nature of the home environment. Respondent rates each eating and activity habit for the participant and both parents as applicable. There are 4 sub-scales: Physical activity, eating habits and style, hunger and satiety cues, and obesogenic environment-exposure.
  Individual scores range from 0 - 4. Sub-scale scores are calculated by summing individual scores in the sub-scale for each family member. A total score was generated by summing all individual scores for each family member. The total score is considered an index of overall inappropriateness of eating patterns, and the higher the score, the more obesogenic the environment.

CONTACTS AND LOCATIONS:
Overall Officials: Amy McPherson, PhD, Principal Investigator — Holland Bloorview Kids Rehabilitation Hospital
Locations (2):
- Canada (2):
  - Thames Valley Children's Centre, London, Ontario
  - Holland Bloorview Kids Rehabilitation Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McPherson AC, Biddiss E, Chen L, Church PT, de Groot JF, Keenan S, King G, Lui T, Maltais DB, Merette C, Moffet H, Moola F, Schwellnus H. Children and Teens in Charge of their Health (CATCH): A protocol for a feasibility randomised controlled trial of solution-focused coaching to foster healthy lifestyles in childhood disability. BMJ Open. 2019 Mar 4;9(3):e025119. doi: 10.1136/bmjopen-2018-025119. PMID 30837255

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-16): https://cdn.clinicaltrials.gov/large-docs/06/NCT03523806/Prot_SAP_000.pdf